CLINICAL TRIAL: NCT03983499
Title: Latinos Understanding the Need for Adherence in Diabetes
Acronym: LUNA-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Gregory Talavera, Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NR014866
Record Dates: First submitted 2019-06-07; First posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Type 2 Diabetes; Glycemic Control; Cardiovascular Risk Factors; Psychological Distress
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Special Intervention (Experimental): The special intervention (SI) arm addresses glycemic control, medication adherence, control of modifiable CVD risk factors, health behavior change, and psychosocial and cultural barriers to self-management. The SI arm consists of a collaborative care team approach with four main elements including: 1) Specialized clinical care by a medical provider; 2) Specialized behavioral health care by a behavioral health provider; 3) Group-based chronic disease self-management education by peer-leaders; 4) Intensive, proactive care coordination facilitated by a patient registry and electronic health records.
  Interventions: Behavioral: Special Intervention
- Usual Care (No Intervention): Participants randomized to the Usual Care (UC) arm continue to see their primary care provider and receive referrals to health education. At the discretion of the provider, UC patients are screened and referred to behavioral health (BH) care.

INTERVENTIONS:
Behavioral: Special Intervention — The components of the Special Intervention (SI) integrated design are: 1) Co-location of the clinical team; 2) Shared medical plan; 3) Clinical visits with a medical provider for management of chronic medical conditions; 4) Visits with behavioral health provider for management of psychosocial chronic conditions; 5) Care coordination; 6) Six group-health education classes and two booster sessions led by a promotora. Participants in the SI arm meet with the integrated care team in the context of a regular medical visit primarily to focus on clinical/biological aspects of the chronic medical conditions (diabetes, dyslipidemia, hypertension, obesity, etc.)
  Other Names: Medical Provider clinical visits; Behavioral Health Provider counseling visits; Care Coordination; Group Health Education
  Arms: Special Intervention

SUMMARY:
The Latinos Understanding the Need for Adherence in Diabetes (LUNA-D) study, is a randomized controlled trial testing the effectiveness of an integrated behavioral health and primary care chronic care disease management intervention for low income Latino patients with type-2 diabetes mellitus (T2DM) that have 2 or more chronic health conditions. LUNA-D focuses on diabetes management and behavioral health care integration.

DETAILED DESCRIPTION:
LUNA-D proposes to test the ability of a fully integrated behavioral health and primary care diabetes management intervention in a federally-qualified community health care setting to improve multiple clinical and behavioral outcomes. LUNA-D will recruit non-insulin using adult type two diabetes mellitus (T2DM) patients with two or more chronic diseases. Half will be randomized to the Special Intervention (SI) arm and half to the Usual Care (UC) arm. The SI is an intensive intervention including fully integrated clinical visits with a medical provider (MP) co-located with a behavioral health counselor (BHC) and peer-led evidence-based group health education sessions and proactive care coordination. Usual Care is represented by passive appointments with the primary care physician and passive referrals to behavioral health and traditional health education. Biological measurements will be taken at baseline, 3-, 6-, 9- and 12-months to detect changes in glycemic control. Clinical lab measures, medication adherence, weight, health behaviors and psychosocial measures will also be obtained across the study.

ELIGIBILITY:
Inclusion Criteria:

This study targets non-insulin using T2DM patients with 2 or more chronic conditions. The primary eligibility criteria are as follows:

* Self-identify as Hispanic/Latino
* Be a registered & established patient of SYH
* 18 years of age or older
* Have an established diagnosis of T2DM (but not currently using insulin)
* Not currently participating in any other diabetes or CVD intervention program
* Have 2 or more CVD risk factors (e.g., depression, anxiety, hypertension, dyslipidemia, obesity, or smoking)

Exclusion Criteria:

Individuals will be excluded if they:

* Are pregnant or planning to get pregnant (temporary exclusion, may qualify 6-months postpartum)
* Have plans to move out of the area in the next 12 months
* Have pre-existing health problems so severe as to prohibit informed consent and study attendance
* Have severe diabetes, including renal disease and/or on dialysis
* Have severe psychosocial conditions under the care of a psychiatrist (e.g., severe depression, bipolar disorder, or schizophrenia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2015-07-16 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
HbA1c Blood Value | Repeated measures will be taken at baseline, 3-, 6-, 9-, 12-months post randomization in order to compare the rates of change over time between the two conditions (SI and UC).
  The primary outcome is change in HbA1c values among non-insulin using type 2 diabetes mellitus Latino patients through a linguistically and culturally appropriate evidence-based application of a Chronic Care Model (LUNA-D).

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Repeated measures will be taken at baseline, 3-, 6-, 9-, 12-months post randomization in order to compare the rates of change over time between the two conditions (SI and UC).
  Lower BMI among non-insulin using type 2 diabetes mellitus Latino patients through a linguistically and culturally appropriate evidence-based application of a Chronic Care Model (LUNA-D).
Total Cholesterol | Repeated measures will be taken at baseline, 3-, 6-, 9-, 12-months post randomization in order to compare the rates of change over time between the two conditions (SI and UC).
  Lower cholesterol levels among non-insulin using type 2 diabetes mellitus Latino patients through a linguistically and culturally appropriate evidence-based application of a Chronic Care Model (LUNA-D).
Blood Pressure (BP) | Repeated measures will be taken at baseline, 3-, 6-, 9-, 12-months post randomization in order to compare the rates of change over time between the two conditions (SI and UC).
  Improve the ratio of systolic to diastolic blood pressure among non-insulin using type 2 diabetes mellitus Latino patients through a linguistically and culturally appropriate evidence-based application of a Chronic Care Model (LUNA-D).
Patient Health Questionnaire (PHQ-8) | Repeated measures will be taken at baseline, 3-, 6-, 9-, 12-months post randomization in order to compare the rates of change over time between the two conditions (SI and UC).
  Improve depression symptomatology among non-insulin using type 2 diabetes mellitus Latino patients through a linguistically and culturally appropriate evidence-based application of a Chronic Care Model (LUNA-D).
Generalized Anxiety Disorder 7-item (GAD-7) | Repeated measures will be taken at baseline, 3-, 6-, 9-, 12-months post randomization in order to compare the rates of change over time between the two conditions (SI and UC).
  Improve anxiety symptomatology among non-insulin using type 2 diabetes mellitus Latino patients through a linguistically and culturally appropriate evidence-based application of a Chronic Care Model (LUNA-D).

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Talavera, MD/MPH, Principal Investigator — SDSU
Locations (1):
- South Bay Latino Research Center, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Castaneda SF, Gallo LC, Garcia ML, Mendoza PM, Gutierrez AP, Lopez-Gurolla M, Roesch S, Pichardo MS, Munoz F, Talavera GA. Effectiveness of an integrated primary care intervention in improving psychosocial outcomes among Latino adults with diabetes: the LUNA-D study. Transl Behav Med. 2022 Aug 17;12(8):825-833. doi: 10.1093/tbm/ibac042. PMID 35776001
- [Derived] Talavera GA, Castaneda SF, Mendoza PM, Lopez-Gurrola M, Roesch S, Pichardo MS, Garcia ML, Munoz F, Gallo LC. Latinos understanding the need for adherence in diabetes (LUNA-D): a randomized controlled trial of an integrated team-based care intervention among Latinos with diabetes. Transl Behav Med. 2021 Sep 15;11(9):1665-1675. doi: 10.1093/tbm/ibab052. PMID 34057186